CLINICAL TRIAL: NCT06242301
Title: Feasibility Assessment of a Collective Person-centered Dialogue (COPE-D) Intervention for Patients Hospitalised with COPD Exacerbation
Brief Title: Is a Collective Person-centered Dialogue Intervention for Hospitalised COPD Patients Feasible?
Acronym: COPE-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Aarhus (Other); Danish Lung Association (Other)
Responsible Party: Principal Investigator, Tanja Sofie Hansen, Principal Investigator, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: COPD dialogue - Feasibility
Record Dates: First submitted 2024-01-14; First posted 2024-02-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: COPD Exacerbation Acute; Nutrition Poor; Physical Inactivity; Relatives
Keywords: COPD; Nutrition; Physical activity; Person-centered; Dialogue
MeSH Terms: conditions — Malnutrition; Sedentary Behavior; Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The COPE-D intervention (Other)
  Interventions: Other: The collective person-centered dialogue intervention

INTERVENTIONS:
Other: The collective person-centered dialogue intervention — * Educate and train the interdisciplinary team and staff.
  * Upon hospitalisation, the interdisciplinary team introduces an interactive dialogue tool to patients and their relatives. The tool is designed to facilitate a person-centered dialogue and assess the patients' needs, motivations, and challenges regarding eating and physical activity during hospitalization and in everyday settings.
  * Following the needs assessment, the interdisciplinary team will introduce and initiate a personalised action plan based on a predefined template that includes suggestions for actions related to the needs assessment.
  * Collaboratively, the interdisciplinary team, patients, and relatives evaluate and adjust the action plan, discussing relevant actions and potential community support for maintaining daily activities.
  * Before discharge, discussions are guided by predefined questions. Patients receive a contact number for follow-up and information on oral nutritional supplementation prescriptions.

SUMMARY:
The aim of this mixed methods trial is to investigate the feasibility of a collective person-centred dialogue (COPE-D) intervention delivered by an interdisciplinary team for a population of patients hospitalised and diagnosed with COPD and their relatives.

The main questions it aims to answer are:

* The clinical uncertainties: What components of the COPE-D intervention are delivered to the included patients? (The data will be collected from the patient's journal record)
* The clinical uncertainties: How acceptable is the COPE-D intervention for the patients, relatives, and the interdisciplinary team? (Answered by patient and relative interviews with a structured interview guide before discharge and 14 days after hospitalisation, and by the interdisciplinary team using focus-group interviews after the intervention enrolment).
* The procedural uncertainties: Are the patients willing to engage in the trial? (Estimated by the inclusion rate).

The interdisciplinary team will be instructed to deliver and document the COPE-D intervention. The primary focus of COPE-D intervention is to prepare and enhance the patient's and relative's ability to regain their everyday life after discharge. The COPE-D intervention includes a dialogue tool based on a needs assessment, an action plan template, and a patient guide that prepares for discharge.

The interdisciplinary team will collaborate with COPD patients and their relatives to:

1. Assess the patient's need for nutrition and physical activity support, both during and after hospitalisation using the dialogue tool.
2. Develop an action plan for nutrition and physical activity support using the action plan template.
3. The interdisciplinary team will provide, adjust, and document the nutritional and physical activity support provided by the action plan.
4. Prior to discharge, patients and their relatives are given a discharge guide with pre-defined questions to ask healthcare professionals, a contact telephone number to the outpatient clinic for follow-up if needed, and information about prescriptions for oral nutritional supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD
* Speak and understand Danish.

Exclusion Criteria:

* Patients in the end-of-life phase.
* Patients living in nursing homes.
* Patients with cognitive impairments avoiding participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Clinical uncertainties - An evaluation of the delivery of the needs assessment and the action plan | Measurements will be taken at one time point for each participant prior to discharge. Measurements will be taken four weeks after the beginning of the intervention.
  Following criteria are considered to evaluate the delivery of the needs assessment and the action plan:
  * If less than 80 % receive the needs assessment based on the dialogue tool or the action plan based on the template, the intervention is considered non-feasible.
  * If 80 to 90 % receive the needs assessment and the action plan, then actions to modify the intervention will be elaborated during the upcoming focus group interview with the interdisciplinary team. Any decision to modify the intervention will be based on the completed analysis of the feasibility.
  * If more than 90 % receive the needs assessment and the action plan, then the delivery is determined as feasible without modifications.
Clinical uncertainties - An evaluation of the delivery of the provision actions provided by the action plan | Measurements will be taken at one time point for each participant prior to discharge. Measurements will be taken four weeks after the beginning of the intervention.
  Following criteria are considered to evaluate the delivery of the provision actions from the action plan:
  * If less than 50 % of the actions planned in the action planner are provided, then the COPD support intervention is considered non-feasible.
  * If less than 75 % of the actions planned in the action planner are provided, then actions to modify the intervention will be elaborated during the upcoming focus group interview.
  The modification of the intervention will be based on the completed feasibility test.
  • If 75 % or above of the actions planned in the action planner are provided, then the COPE-D intervention is considered feasible without modifications.
Clinical uncertainties - An evaluation of the patients and their relative acceptability of the intervention. | Measurements will be taken at one time point for each participant prior to discharge. Measurements will be taken four weeks after the beginning of the intervention.
  Following criteria are considered to evaluate the patients and their relative acceptability of the intervention.
  * If less than 50 % of the patient responses contain a positive prompt, then the intervention is considered non-feasible.
  * If between 50- 75 % of the patient responses contain a positive prompt, then actions to modify the intervention will be elaborated during the upcoming focus group interview.
  Any decision to modify the intervention will be based on the completed analysis of the feasibility.
  • If 75 % or above of the patient responses contain a positive prompt, then the COPE-D intervention is considered feasible without modifications.
Clinical uncertainties - An evaluation of the interdisciplinary team members acceptability of the intervention | The measurement will be assessed after the intervention at week six
  The assessment will be measured qualitatively. Focus group interviews will be conducted using a semi-structured interview guide.
Procedural uncertainties - An evaluation of the patients willingness to participate | .Measurement will be taken during recruitment. Measurements will be taken four weeks after the beginning of the intervention.
  Following criteria are considered to evaluate the recruitment for paricipation in the intervention:
  * If less than 30% are willing to participate in the intervention, then the intervention is considered not feasible.
  * If recruitment falls within the range of 30% to 75%, modifications will be considered.
  Determine contextual factors that may influence the recruitment process. Discuss in the focus group interviews with the interdisciplinary team and with the department managers about potential contextual factors that may influence the low recruitment rate.
  • If 75% or more are recruited, the study is deemed feasible without modifications.

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Sofie Hansen, MScN, Principal Investigator — Region h; Ingrid Poulsen, Prof., Study Chair — Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital, Amager, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No